CLINICAL TRIAL: NCT04470531
Title: Role of Co-trimoxazole in Severe COVID-19 Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Collaborators: Anwar Khan Mordern Medical College and Hospital, Dhaka (Unknown); Mugda Medical College and Hospital, Dhaka (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Shohael Mahmud Arafat, Chairman and professor of internal medicine, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2020/6969
Record Dates: First submitted 2020-07-11; First posted 2020-07-14 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Covid19; Severe COVID-19 Patients
MeSH Terms: conditions — COVID-19 | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Intervention Model Description: Arm A :control group will receive standard treatment, Arm B: experimental group will receive standard care and oral co-triamoxazole
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Arm A :No Intervention/control: Standard treatment
  1. Antibiotics for secondary bacterial infection as per institutional guidelines
  2. Supplemental oxygen (to keep saturations between 90% to 96%)
  3. Intravenous hydration (to maintain euvolumia)
  4. Thrombo-prophylaxis as per local guidelines
  5. Paracetamol (oral or I/V 1gram QDS as required or regular)
  6. To consider steroids if indicated (i.e. acute exacerbation of COPD or acute severe asthma)
- intervention /experimental (Experimental): Arm B: Experimental Arm received oral co-trimoxazole + standard therapy
  The following treatments are recommended as standard therapy:
  1. Antibiotics for secondary bacterial infection as per institutional guidelines
  2. Supplemental oxygen (to keep saturations between 90% to 96%)
  3. Intravenous hydration (to maintain euvolumia)
  4. Thrombo-prophylaxis as per local guidelines
  5. Paracetamol (oral or I/V 1gram QDS as required or regular)
  6. To consider steroids if indicated (i.e. acute exacerbation of COPD or acute severe asthma)
  Interventions: Drug: oral co-trimoxazole

INTERVENTIONS:
Drug: oral co-trimoxazole — oral co-trimoxazole + standard therapy
  Other Names: co-trimoxazole
  Arms: intervention /experimental

SUMMARY:
Coronavirus Disease 19 (COVID-19) is a global pandemic caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Severe disease occurs in 15% of the cases with COVID-19 and may progress to critical disease in only 5% of the cases with a high risk of mortality. Critical disease may present as acute respiratory failure secondary to Acute Respiratory Distress Syndrome (ARDS) and is caused by the body's hyper-immune response to the virus in the form of a cytokine storm syndrome (CSS). There is currently no effective anti-viral treatment against SARS-CoV-2 and the mainstay of treatment is supportive. Co-trimoxazole (combination of trimethoprim and sulphamethoxazole in a 1:5) ratio is a Sulphur containing anti-folate bactericidal antibiotic indicated for the treatment of respiratory tract infections. It has been around for over 60 years and is inexpensive and readily available with a good safety profile. It has a rapid onset of action with excellent bioavailability and lung penetration. In addition to having antimicrobial properties co-trimoxazole have immunomodulatory and anti-inflammatory properties and may be a potential treatment option for cytokine storm syndrome mediated severe COVID-19.

This open-label randomized controlled trial will be conducted in the department of medicine at Bangabandhu Sheikh Mujib Medical University (BSMMU), Anwar Khan Modern Medical college and Mughda Medical College Hospital (DMCH), Dhaka for a duration of 6 months following approval of this protocol. It will recruit at least 94 consecutive adults (18 years or older) patients with clinically suspected COVID-19 and severe illness as per WHO criteria. After taking informed written consent patients will be randomly assigned in a 1:1 ratio to either oral co-trimoxazole in addition to standard therapy or standard therapy alone. Baseline characteristics, changes in the physiological and biochemical parameters like (SpO2/FiO2 ratio, respiratory rate, body temperature and C - reactive protein), length of hospital stay, side effects of drugs, requirement for ventilatory support (non-invasive and invasive ventilation) and in-patient mortality between the two groups will be compared.

Conclusion If the results from this clinical trial demonstrate the beneficial effects of co-trimoxazole in severe COVID-19 patients it could be used widely, thereby reducing the need for respiratory support and potentially saving thousands of lives in developing nations with limited resources where healthcare may be easily overwhelmed.

DETAILED DESCRIPTION:
Coronavirus disease (COVID-19) caused by SARS-COV2, represents a highly transmissible and potentially fatal disease that is of great global public health concern at this moment. The pandemic situation in Bangladesh is also evolving rapidly with positive cases and deaths increasing each day. Epidemiological changes in COVID-19 infection should be monitored taking into account potential routes of transmission and subclinical infections, in addition to the adaptation, evolution, and virus spread among humans and possible intermediate animals and reservoirs. But till today there is no specific management to deal with this highly deadly viral infection. Howeverthere are few drugs which might cause some beneficial effects in the recovery of the patient. Cotrimoxazole is a time tested antibiotic which has been in clinical use for 60 years with anti-bacterial action against a wide range of organism. In addition to the antimicrobial effects, co-trimoxazole has anti-inflammatory and immunomodulatory effects. Co-trimoxazole has previously been shown to exert anti-cytokine effect by inhibiting interleukin 1, 6 (IL-1, IL-6) and Tumour Necrosis Factor α (TNF α) which are the major cytokines identified in patients with severe COVID-19. As in some case reports this has shown significant clinical improvement in ARDS, so there is a possibility, that cotrimoxazole might have also role in improving the clinical outcome in COVID-19 patients especially in moderate to severe cases. As till today there is no specific treatment for COVID-19 infections, if cotrimoxazole ifs found to be effective this will bring a great benefit to the target populations. Beside this, cotrimoxazole is a very cheap drug in comparison to other ones this will also be of great economical benefit in taking cares of the general population. As there is no such study published about the role of cotrimoxazole in COVID-19 patients, this study will generate a new information which bring a great benefit in battling with the COVID-19 infection.

Research Question:

What is the outcome of co-trimoxazole in severe COVID-19 patients?

Objectives:

General Objectives To assess the clinical outcome of co-trimoxazolein patients with severe COVID-19

Specific Objectives:

To assess length of stay who are treated with co-trimoxazole in addition to standard treatment versus standard treatment alone.

To find out side effects (rash.itching. dizziness, headache, nausea,vomiting, diarrhea, sore throat, unusual bruising or bleeding, yellowing of the skin or eye discolorations, joint or muscle pain,red or purple skin.etc) of drugs who are treated with co-trimoxazole in addition to standard treatment versus standard treatment alone.

To find out requirement for ventilator support (non-invasive and invasive ventilation) who are treated with co-trimoxazole in addition to standard treatment versus standard treatment alone.

To assess the mortality in patients with severe COVID-19 who are treated with co-trimoxazole in addition to standard treatment versus standard treatment alone.

Study design:Open-label randomized controlled trial Study duration: Six months.

Study Population:

Patients presenting to participating hospitals in Bangladesh with symptoms ofCOVID-19 will be assessed for eligibility.

Inclusion criteria

1. Diagnosed COVID-19 patients ( RT-PCR positive for COVID-19)
2. Age > 18 years
3. Hypoxic respiratory failure (saturation <90% on air at rest or increasing oxygen requirement)
4. Chest examination findings of bilateral crackles on auscultation or chest x-ray showing bilateral infiltrates
5. C-Reactive Protein > 50mg/L

Exclusion criteria

1. Multi-organ failure
2. Severe ARDS (requiring ventilator support on presentation in the form of invasive or non-invasive ventilation)
3. Septic Shock
4. Severe liver disease
5. Acute Kidney Injury (where GFR< 15 and plasma-sulfamethoxazoleconcentration cannot be monitored)
6. Drug allergy/intolerance to co-trimoxazole / Sulphar sensitivity
7. Pregnancy
8. Already receiving Tocilizumab or convalescent therapy Sampling procedure:This RCT will consist of two arms, experimental group and control group.Randomized (1:1) case: control, (non-blinded) trial.

   1. control group will receive standard treatment,
   2. experimental group will recivestandard care and oral co-triamoxazole. Forty-seven (47) patients will be enrolled for each arm. Randomization will be done by a random number table. Allocations will be in sequentially numbered.

Treatment protocol Eligible patients will be received either to oral co-trimoxazole + standard therapy or standard therapy alone. (According to institution /national protocol)

The following treatments are recommended as standard therapy:

1. Antibiotics for secondary bacterial infection as per institutional guidelines
2. Supplemental oxygen (to keep saturations between 90% to 96%)
3. Intravenous hydration (to maintain euvolumia)
4. Thrombo-prophylaxis as per local guidelines
5. Paracetamol (oral or I/V 1gram QDS as required or regular)
6. To consider steroids if indicated (i.e. acute exacerbation of COPD or acute severe asthma) NOTE: The dose of co-trimoxazoleis 960 mg (trimethoprim 160mg + sulphamethoxazole 800mg) twice daily for 7 days orally.

sample size: 94

Research instrument:

1. General questionnaire for assessing socio-demographic data.
2. A checklist of clinical findings
3. A checklist of investigation findings.

Measures Variable:

Data collection required for both groups (co-trimoxazole + standard therapyand standard therapy alone)

1. Age
2. Sex
3. Ethnicity
4. Past medical history - Hypertension, use of ACEI or ARB, DM, IHD, COPD, CKD, Obesity (BMI) andCancer
5. Presenting symptoms (dry cough, productive cough, fever, sore throat, myalgia, lethargy, headache, breathlessness, nausea, diarrhoea and any other)
6. Baseline observations on dayof initiating treatment (Day 0): oxygen saturation(SpO2), fraction of inspired oxygen (FiO2) , SpO2/FiO2 ratio, respiratory rate, body temperature, neutrophil-lymphocyte ratio, C-Reactive Protein&findings of bilateral infiltrates on chest-x-ray.
7. Follow-up observations after randomization on Day 1,2,3,4 and 5 for SpO2/FiO2 ratio, respiratory rate,body temperature and C-Reactive Protein
8. Length of stay (in days)
9. Use of ventilator support (invasive or non-invasive ventilation)
10. Side effects of drugs
11. In-patient mortality Primary end points

1. Length of stay in hospital (in days) 2. In-patient mortality

Secondary end points

1. Change in observations after randomization on Day 1,2,3,4 and 5 for SpO2/FiO2 ratio, respiratory rate, body temperature and C-Reactive Protein
2. Use of ventilator support (invasive or non-invasive ventilation)
3. Side effects of drugs co-trimoxazole

Data Collection procedure:

Pre-designed case record form (CRF) will be used for collecting data, which will also contain the result of the study. The information collected in the CRF will be reviewed and inconsistencies will be investigated and clarified. Data from case record forms will be anonymised and stored securely in a secure online web-based portal.

Statistical analysis: Statistical analysis will be performed using t-test or Mann -Whitney U test or Wilcoxon signed rank test for continuous variables and Chi- square test or Fisher's exact test for categorical variables. Survival will be assessed by the Kaplan-Meier method. Comparisons between two groups will be performed using the log-rank test and Hazard regression test.A p-value of < 0.05 will be considered to be significant. The statistical software SPSS version 25 will be used for the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed COVID-19 patients ( RT-PCR positive for COVID-19)
2. Age > 18 years
3. Hypoxic respiratory failure (saturation <90% on air at rest or increasing oxygen requirement)
4. Chest examination findings of bilateral crackles on auscultation or chest x-ray showing bilateral infiltrates
5. C-Reactive Protein > 50mg/L

Exclusion Criteria:

1. Multi-organ failure
2. Severe ARDS (requiring ventilator support on presentation in the form of invasive or non-invasive ventilation)
3. Septic Shock
4. Severe liver disease
5. Acute Kidney Injury (where GFR< 15 and plasma-sulfamethoxazoleconcentration cannot be monitored)
6. Drug allergy/intolerance to co-trimoxazole / Sulphar sensitivity
7. Pregnancy
8. Already receiving Tocilizumab or convalescent therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2020-07-12 (Actual); Primary Completion 2020-10-12 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Length of stay in hospital (in days) | 14 days
  Duration of hospital stay in days
In-patient mortality | 14 days
  % of patients died after enrollment

SECONDARY OUTCOMES:
SpO2/FiO2 ratio | Day 1,2,3,4 and 5
  ratio of Saturation of oxygen in % and Fraction of inspired oxygen
respiratory rate | Day 1,2,3,4 and 5
  Respiratory rate per minute
C-reactive Protein | Day 1,2,3,4 and 5
  CRP level in mg/litre
Fever | Day 1,2,3,4 and 5
  Temperature in degree Fahrenheit
Ventilator support | 14 days
  Requirement of ventilator support in hours
Proportion of drug adverse reaction | 24 hours
  % of patients developed early reaction like fever, rash, abdominal pain, urticaria, vomiting, wheezing, chest tightness

CONTACTS AND LOCATIONS:
Overall Officials: Shohael Arafat, Study Chair — ICMJE
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the journal authority and make public as part of the publication
Supporting Information: SAP, ICF, CSR
Time Frame: six months
Access Criteria: Available on public domain like figshare, researchgate and others